CLINICAL TRIAL: NCT05246111
Title: Phase I Study to Evaluate the Mass Balance, PK, Metabolism and Excretion of Berzosertib (Intravenous) Containing Microtracer [14C]Berzosertib in Participants With Advanced Solid Tumors (DDRiver Solid Tumors 208)
Brief Title: Berzosertib Human Mass Balance Study (DDRiver Solid Tumors 208)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS201923_0008; 2021-002226-24 (EudraCT Number)
Record Dates: First submitted 2022-01-13; First posted 2022-02-18 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor
Keywords: Topotecan; Ataxia telangiectasia mutated and Rad3-related (ATR) protein; ATR inhibitor; M6620; Berzosertib; Mass balance
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — berzosertib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [14C]Berzosertib (Experimental): Participants received single intravenous infusion of[14C]Berzosertib at a dose of 210 milligrams per square meter (mg/m^2) on Day 1 in Period 1 and stay in clinical research unit (CRU) is required until the discharge criteria are met with a maximum confinement period of 15 days.
  Interventions: Drug: [14C]Berzosertib
- Berzosertib + Topotecan (Experimental): Participants received single intravenous infusion of Berzosertib at a dose of 210 mg/m^2 on Day 2 and Day 5 in combination with topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in period 2 until disease progression or other criteria for study intervention discontinuation were met.
  Interventions: Drug: Berzosertib; Drug: Topotecan

INTERVENTIONS:
Drug: [14C]Berzosertib — Participants received single intravenous infusion of [14C]Berzosertib at a dose of 210 milligrams per square meter (mg/m^2) on Day 1 in Period 1 and stay in clinical research unit (CRU) is required until the discharge criteria are met with a maximum confinement period of 15 days.
  Other Names: M6620
  Arms: [14C]Berzosertib
Drug: Berzosertib — Participants received single intravenous infusion of Berzosertib at a dose of 210 mg/m^2 on Day 2 and Day 5 in period 2 until disease progression or other criteria for study intervention discontinuation were met.
  Other Names: M6620
  Arms: Berzosertib + Topotecan
Drug: Topotecan — Participants received topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle in period 2 until disease progression or other criteria for study intervention discontinuation were met.
  Arms: Berzosertib + Topotecan

SUMMARY:
The study was conducted in two periods, Period 1 (mass balance) and Period 2 (extension). The purpose of Period 1 of this study was to provide a quantitative characterization of the mass balance, rates and routes of elimination, and metabolic pathways after a single intravenous administration of [14C]berzosertib. The purpose of Period 2 was to assess safety and efficacy of berzosertib in combination with topotecan.

ELIGIBILITY:
Inclusion Criteria: .

* Histologically proven advanced solid tumors that are considered appropriate for treatment in Period 2 of this study, for which no effective standard therapy exists, or standard therapy has failed or cannot be tolerated
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) =< 1
* Evaluable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) at Screening
* Participant has adequate renal, hematological and hepatic function
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with uncontrolled intercurrent illness including, but not limited to, severe active infection including, acute respiratory syndrome coronavirus-2 infection/coronavirus disease 2019 (Covid 19), immune deficiencies, uncontrolled diabetes, uncontrolled arterial hypertension and symptomatic congestive heart failure
* Concurrent participation in another interventional clinical study is not permitted.
* Known hypersensitivity to the study interventions, a similar structural compound, or to one or more excipients used
* Prior or concurrent treatment with a nonpermitted drug/intervention from the first dose of study intervention administration, as defined per protocol.
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (2):
- Hungary (2):
  - Magyar Honvédség Egészségügyi Központ, Podmaniczky utcai telephely, Onkológiai Osztály, Budapest
  - PRA Magyarország Kft. Fázis I-es Klinikai Farmakológiai Vizsgálóhely, Budapest

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201923_0008
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: DDRiver website — http://www.DDRiver-trials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First Participant Signed Informed Consent: 15-Feb-2022; Last Participant Last Visit: 28-Jun-2023
Period: Period 01
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan
Started | 6 | 0
Completed | 5 | 0
Not Completed | 1 | 0
Not completed — NOT ELIGIBLE IC5 | 1 | 0
Period: Period 02
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan
Started | 0 | 5 (Only 5 participants rolled over to Period 2.)
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants received single intravenous infusion of [14C]Berzosertib at a dose of 210 milligrams per square meter (mg/m^2) on Day 1 in Period 1 and stay in clinical research unit (CRU) is required until the discharge criteria are met with a maximum confinement period of 15 days. In Period 2, participants received single intravenous infusion of Berzosertib at a dose of 210 mg/m^2 on Day 2 and Day 5 in combination with topotecan at a dose of 1.25 mg/m^2 intravenously on Days 1 through 5 of each 21-day cycle until disease progression or other criteria for study intervention discontinuation were met.
Arm/Group | All Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Percent Urinary Recovery (Feurine) of Total Radioactivity
Description: Feurine, fractions of total radioactivity excreted in urine as percentage of the administered dose between time t1 (= start) and t2 (= end).
Time Frame: Predose, 0-4, 4-12, 12-24, 24-48, 48-72, 72-96, 96-120, 120-144 and 144-168 hours after dosing on Day 1, continued in 24-hour intervals, until discharge criteria are met, assessed up to Day 14 post-dose
Population: The Pharmacokinetic (PK) Analysis Set was a subset of the safety analysis set (SAF) included all participants who received at least one dose of Investigational Manufacturing product (IMP), in Period 1 and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of administered dose (%)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
percentage of administered dose (%) | 15.8 (3.2)

2. Primary Outcome: Period 1: Percent Fecal Recovery (Fefeces) of Total Radioactivity
Description: Fefeces, fractions of total radioactivity excreted in feces as percentage of the administered dose between time t1 (= start) and t2 (= end).
Time Frame: as for outcome 1
Population: PK Analysis Set was a subset of the SAF included all participants who received at least one dose of IMP, in Period 1 and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of administered dose (%)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
percentage of administered dose (%) | 73.7 (6.56)

3. Primary Outcome: Period 1: Percent Total Recovery in Urine and Feces (Fetotal) of Total Radioactivity
Description: Fetotal, fractions of total radioactivity excreted in urine and feces as percentage of the administered dose between time t1 (= start) and t2 (= end).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of administered dose (%)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
percentage of administered dose (%) | 89.5 (7.04)

4. Primary Outcome: Period 1: Maximum Observed Plasma Concentration (Cmax) of Berzosertib
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours after dosing on Day 1, continued in 24-hour intervals, until discharge criteria are met, assessed up to Day 14 post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL) | 1870 (12.7)

5. Primary Outcome: Period 1: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Berzosertib
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
hour*nanogram per milliliter (h*ng/mL) | 8620 (23.0)

6. Primary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Berzosertib
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Lambda z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration is at or above the Lower Limit of quantification (LLOQ) and Lambda z was the apparent terminal rate constant determined by log-linear regression analysis of the measured plasma concentrations of the terminal log-linear phase.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
h*ng/mL | 8650 (23.0)

7. Primary Outcome: Period 1: Terminal Elimination Half-Life (T1/2) of Berzosertib
Description: Elimination Half Life (T1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half. T1/2 was calculated by natural log 2 divided by Lambda z. Lambda z was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
hours | 19.6 (19.9)

8. Primary Outcome: Period 1: Total Body Clearance (CL) of Berzosertib From Plasma
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body, calculated as dose divided by AUC0-infinity.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
liter per hour | 47.7 (32.7)

9. Primary Outcome: Period 1: Apparent Volume of Distribution During the Terminal Phase (Vz) of Berzosertib
Description: Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz = Dose/AUC0-inf multiply Lambda z.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
liters | 1340 (31.1)

10. Primary Outcome: Period 1: Apparent Volume of Distribution at Steady State (Vss) of Berzosertib
Description: Vss is the theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it is in blood plasma at steady state.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
liters | 930 (24.7)

11. Primary Outcome: Period 1: Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity
Description: Cmax was obtained directly from the plasma concentration versus time curve. Cmax of total radioactivity was calculated in nanogram equivalents per milliliter (ng eq)/mL.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng eq)/mL
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
(ng eq)/mL | 2410 (19.2)

12. Primary Outcome: Period 1: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Total Radioactivity
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule. AUC0-t was calculated in hour*nanogram equivalents per milliliter (h*[ng eq/mL]).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng eq/mL
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
h*ng eq/mL | 38300 (19.0)

13. Primary Outcome: Period 1: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Total Radioactivity
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng eq/mL
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
h*ng eq/mL | 39400 (19.2)

14. Primary Outcome: Period 1: Terminal Elimination Half-Life (T1/2) of Total Radioactivity
Description: as for outcome 7
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
hours | 64.3 (30.1)

15. Primary Outcome: Period 1: Maximum Observed Blood Concentration (Cmax) of Total Radioactivity
Description: Cmax was obtained directly from the blood concentration versus time curve.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
ng eq/mL | 2920 (9.7)

16. Primary Outcome: Period 1: Area Under the Blood Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Total Radioactivity
Description: Area under the blood concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(ng eq/mL)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
h*(ng eq/mL) | 33100 (23.8)

17. Primary Outcome: Period 1: Area Under the Blood Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Total Radioactivity
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*(ng eq/mL)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
h*(ng eq/mL) | 33900 (23.1)

18. Primary Outcome: Period 1: Terminal Elimination Half-Life (T1/2) of Total Radioactivity in Blood
Description: as for outcome 7
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
hours | 30.6 (50.6)

19. Primary Outcome: Period 1: Cumulative Amount of Berzosertib Dose Excreted in Urine (Aeurine)
Description: Aeurine is defined as the amount of Berzosertib excreted in urine over the time interval from t1 (= start) and t2 (= end).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram equivalent (mg eq)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
milligram equivalent (mg eq) | 41.1 (14.8)

20. Primary Outcome: Period 1: Percentage of Berzosertib Dose Excreted in Urine (Feurine)
Description: Feurine is defined as the amount of Berzosertib unchanged excreted in urine as percentage of the administered dose over the time interval t1 (= start) and t2 (= end).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of administered dose (%)
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
percentage of administered dose (%) | 9.84 (2.74)

21. Primary Outcome: Period 1: Renal Clearance (CLr) of Berzosertib
Description: Renal clearance was calculated as total amount of unchanged drug excreted in the urine between times t1 and t2 (Aeurine) divided by area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | [14C]Berzosertib
Number analyzed (Participants) | 5
liter per hour | 7.84 (2.86)

22. Secondary Outcome: Period 1 and Period 2: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, heart rate, systolic and diastolic blood pressure and respiration rate. Number of participants with clinically significant findings in vital signs were reported. Clinical significance was decided by Investigator.
Time Frame: Period 1: Baseline up to Day 14; Period 2: From Day 1 of period 2 until disease progression or other criteria for study intervention discontinuation are met (up to a maximum of approximately 16 months)
Population: SAF included all participants who had received any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

23. Secondary Outcome: Period 1 and Period 2: Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Measurements
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. 12-lead ECG recordings were obtained after the participants have rested for at least 10 minutes in semi-supine position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: as for outcome 22
Population: SAF included all participants who had received any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

24. Secondary Outcome: Period 1 and Period 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment Related TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal relationship with this treatment. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, regardless if it is considered related to the medicinal product. Serious AE: AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs are defined as AEs that were reported or worsened on or after start of study drug dosing through the Safety Follow-up Visit. TEAEs included both serious TEAEs and non-serious TEAEs. Treatment related AEs: reasonably related to the study drug/study treatment.
Time Frame: as for outcome 22
Population: SAF included all participants who had received any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan
Number analyzed (Participants) | 6 | 5
Participants
  TEAEs | 6 | 5
  Treatment Related TEAEs | 4 | 5

ADVERSE EVENTS:
Time Frame: Period 1: Baseline up to Day 14; Period 2: From Day 1 of period 2 until disease progression or other criteria for study intervention discontinuation are met, assessed up to 16 months
Arm/Group | [14C]Berzosertib | Berzosertib + Topotecan | All Participants
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/5 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/5 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]Berzosertib (N=6) | Berzosertib + Topotecan (N=5) | All Participants (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]Berzosertib (N=6) | Berzosertib + Topotecan (N=5) | All Participants (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 3 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (9) | 3 (9)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 4 (4) | 0 (0) | 4 (4)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Transfusion related complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT05246111/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT05246111/SAP_001.pdf